CLINICAL TRIAL: NCT02990247
Title: Home Telemonitoring of Resting Spontaneous Breathing in Severe Asthma: a Pilot Study
Acronym: AsthmaDom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CHUBX 2015/04
Record Dates: First submitted 2016-12-02; First posted 2016-12-13 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Asthma
Keywords: Asthma; Exacerbations; Telemonitoring; Biomarkers
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AMARS (Experimental): Evaluation the resting ventilatory flow by applying a new technique called anharmonic morphological analysis of the respiratory signals (AMARS).
  Interventions: Device: anharmonic morphological analysis of the respiratory signals (AMARS)

INTERVENTIONS:
Device: anharmonic morphological analysis of the respiratory signals (AMARS)

SUMMARY:
Asthma exacerbations account for a significant morbidity and disproportionate health care costs. However, there is no currently available biomarker or lung function parameter that can accurately predict the risk of future exacerbations. The current work aims at evaluating the resting ventilatory flow by applying a new technique called anharmonic morphological analysis of the respiratory signals (AMARS). We hypothesize that monitoring AMARS is potentially able to detect an increased risk of asthma exacerbations.

DETAILED DESCRIPTION:
Asthma exacerbations represent an acute or sub-acute worsening in symptoms and lung function from the patient's usual status. Early detection of exacerbations is a major public health issue. In clinic, management of asthma involves asthma control questionnaires and pulmonary function tests (Forced Expiratory Volume (FEV1), Fractional exhaled nitric oxide or FeNO). At home, the peak expiratory flow rate (PEFR) measured by the peak flow meter is an aid to monitor asthma but its ability to predict asthma exacerbations remains controversial. Anharmonic morphological analysis of the respiratory signals (AMARS) is a new morpho-mathematic biomarker that produces objective and accurate measures of the shape of the ventilatory flow. The current study aims at monitoring the resting spontaneous breathing at home in asthmatics. Changes in AMARS may be a predictor of early symptoms of asthma exacerbations. We will recruit 120 asthmatic patients. Patients will be given a portable device for telemonitoring. Resting spontaneous breathing will be measured during 2-3 min in the morning and in the evening, twice a week at least for 12 months. Three visits will be scheduled in Clinical Investigation Center before (V1), after 6-month (V2) and 12-month (V3) telemonitoring period.

ELIGIBILITY:
Inclusion Criteria:

* male or female aged more than 18 yrs
* written informed consent
* diagnosis of asthma according to Global Initiative For Asthma (GINA) criteria
* history of at least one moderate to severe exacerbation in the previous 12 months

Exclusion Criteria:

* smoker or former smoker (> 10 packs-year)
* concomitant asthma exacerbation (at V1)
* prisoners
* protected adults
* no affiliation to the French Social Security System

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2018-11-06 (Actual); Study Completion 2018-11-06 (Actual)

PRIMARY OUTCOMES:
Sensibility parameters resting breath parameter to predict asthma exacerbation | 12 months
Specificity of resting breath parameters to predict asthma exacerbation | 12 months
Positive predictive value of resting breath parameters to predict asthma exacerbation | 12 months
Negative predictive value of resting breath parameters to predict asthma exacerbation | 12 months

SECONDARY OUTCOMES:
FEV1 | Day 1
  Volume that has been exhaled at the end of the first second of forced expiration
FEV1 | 6 months
  Volume that has been exhaled at the end of the first second of forced expiration
FEV1 | 12 months
  Volume that has been exhaled at the end of the first second of forced expiration
Asthma exacerbation severity | Day 1
  The number of asthma exacerbations between Day 1 and month 12 will be quoted and defined according to the protocol (abnormal asthma symptoms increase requiring change in asthma medication). Each exacerbation will be quoted according to its severity as mild (requiring increased in inhaled beta2 agonists use for 7 days as assessed by item6 of the Asthma Control Questionnaire (ACQ)), moderate (requiring short course of oral steroid and/or antibiotics) or severe (i.e., requiring hospitalization).
Asthma exacerbation severity | 12 months
  The number of asthma exacerbations between Day 1 and month 12 will be quoted and defined according to the protocol (abnormal asthma symptoms increase requiring change in asthma medication). Each exacerbation will be quoted according to its severity as mild (requiring increased in inhaled beta2 agonists use for 7 days as assessed by item6 of the Asthma Control Questionnaire (ACQ)), moderate (requiring short course of oral steroid and/or antibiotics) or severe (i.e., requiring hospitalization).
Asthma quality of life questionnaires | Day 1
Asthma quality of life questionnaires | 6 months
Asthma quality of life questionnaires | 12 months
Asthma Control Test questionnaires | day 1
Asthma Control Test questionnaires | 6 months
Asthma Control Test questionnaires | 12 months
Forced Vital Capacity (FVC) | day 1
  Forced vital capacity: the determination of the vital capacity from a maximally forced expiratory effort
FVC | 6 months
  Forced vital capacity: the determination of the vital capacity from a maximally forced expiratory effort
FVC | 12 months
  Forced vital capacity: the determination of the vital capacity from a maximally forced expiratory effort
FEV1/FVC ratio | Day 1
FEV1/FVC ratio | 6 months
FEV1/FVC ratio | 12 months
Forced Expiratory Flow (FEF25-75%) | Day 1
  Forced expiratory flow related to some portion of the FVC curve; modifiers refer to amount of FVC already exhaled
FEF25-75% | 6 months
  Forced expiratory flow related to some portion of the FVC curve; modifiers refer to amount of FVC already exhaled
FEF25-75% | 12 months
  Forced expiratory flow related to some portion of the FVC curve; modifiers refer to amount of FVC already exhaled
PEF | Day 1
  Peak expiratory flow: The highest forced expiratory flow measured with a peak flow meter
PEF | 6 months
  Peak expiratory flow: The highest forced expiratory flow measured with a peak flow meter
PEF | 12 months
  Peak expiratory flow: The highest forced expiratory flow measured with a peak flow meter

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Berger, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (2):
- France (2):
  - Grenoble University Hospital, Grenoble
  - Bordeaux University Hospital, Pessac

IPD SHARING:
Plan to Share IPD: No